CLINICAL TRIAL: NCT06397001
Title: An Open-label Single Center, Single Patient Study of an Experimental Antisense Oligonucleotide (ASO) Treatment in AA Amyloidosis
Brief Title: Treatment of AA Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nelson Leung, MD (Other)
Responsible Party: Sponsor-Investigator, Nelson Leung, MD, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-005092
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: AA Amyloidosis
MeSH Terms: conditions — AA amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nL-SAA1-01 (Experimental): Subject will receive subcutaneous injection of nL-SAA1-01
  Interventions: Drug: nL-SAA1-01

INTERVENTIONS:
Drug: nL-SAA1-01 — Personalized antisense oligonucleotide

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a subcutaneous injection of nL-SAA1-01in a patient with AA Amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven AA amyloidosis
* Measurable disease
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records

Exclusion Criteria:

* Participant has any condition that in the opinion of the site investigator, would ultimately prevent the completion of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events and/or serious adverse events | 1 year
  Number of adverse events and/or serious adverse events experienced

SECONDARY OUTCOMES:
Change in kidney function | Baseline, 1 year
  The change in kidney function is measured by the glomerular filtration rate (GFR)
Change in quality of life - physical well-being | Baseline, 1 year
  Physical well-being will be measured using a Linear Analog Scale Assessment (LASA) The Likert scale runs from 0 (as bad as possible) to 10 (as good as possible) where a higher rating suggest a higher quality of life.
Change in quality of life - emotional well-being | Baseline, 1 year
  Emotional well-being will be measured using a Linear Analog Scale Assessment (LASA) The Likert scale runs from 0 (as bad as possible) to 10 (as good as possible) where a higher rating suggest a higher quality of life.
Change in quality of life - spiritual well-being | Baseline, 1 year
  Spiritual well-being will be measured using a Linear Analog Scale Assessment (LASA) The Likert scale runs from 0 (as bad as possible) to 10 (as good as possible) where a higher rating suggest a higher quality of life.
Change in quality of life - intellectual well-being | Baseline, 1 year
  Intellectual well-being will be measured using a Linear Analog Scale Assessment (LASA) The Likert scale runs from 0 (as bad as possible) to 10 (as good as possible) where a higher rating suggest a higher quality of life.
Change in quality of life - overall well-being | Baseline, 1 year
  Overall well-being will be measured using a Linear Analog Scale Assessment (LASA) The Likert scale runs from 0 (as bad as possible) to 10 (as good as possible) where a higher rating suggest a higher quality of life.
Initiation of dialysis | 1 year
  The amount of time between the first dose of the investigational product and the need for dialysis
Initiation of kidney transplantation | 1 year
  The amount of time between the first dose of the investigational product and the need for a kidney transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Leung, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No